CLINICAL TRIAL: NCT05460338
Title: Effect of Oral Vitamin D on Oxidative Stress and Inflammation in Hemodialysis
Brief Title: Vitamin D, Oxidative Stress and Inflammation in Hemodialysis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona AlShahawey Ghazy, PhD, Assistant professor of Clinical Pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PhCl37
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Oxidative Stress; Inflammation; Vitamin D Deficiency
MeSH Terms: conditions — Inflammation; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly Cholecalciferol Group (Active Comparator): 25 hemodialysis patients on oral cholecalciferol 50.000IU Cholecalciferol, once weekly, taken post-hemodialysis session for 3 months.
  Interventions: Drug: Cholecalciferol
- Monthly Cholecalciferol Group (Active Comparator): 25 hemodialysis patients on Oral 200.000IU Cholecalciferol, once monthly, for 3 months.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — native form of Vitamin D.

SUMMARY:
Vitamin D deficiency is now considered a global problem in general population, but it seemed to be more prominent in chronic kidney disease (CKD) patients, especially those on regular hemodialysis. Being a key regulator in mineral metabolism, there's also emerging evidences linking vitamin D deficiency with inflammation and oxidative stress, which are both recognized as constant threats to cardiovascular outcomes in hemodialysis patients.

It's prospective, randomized trial that's carried out to evaluate the effect of weekly versus, monthly oral cholecalciferol, on vitamin D (25(OH)D) levels, oxidative stress markers, inflammatory markers and secondary hyperparathyroidism in hemodialysis patients. Fifty eligible hemodialysis patients were randomly assigned to either Group A (Oral 50.000IU Cholecalciferol, once weekly) or Group B (Oral 200.000IU Cholecalciferol, once monthly), for 3 months. Serum levels of (25(OH)D), serum malondialdehyde (MDA), serum superoxide dismutase (SOD), serum high sensitive (hsCRP), calcium, phosphorus, and intact parathormone (iPTH) levels, were all assessed at baseline and at the end of the study

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18-70 years, on maintenance hemodialysis for a duration of 3 months or more, in a stable clinical condition (no hospitalization in the previous 3 months), with serum vitamin D levels of < 30 ng/ml.

Exclusion Criteria:

* Patients with hypersensitivity to cholecalciferol, ongoing cholecalciferol therapy, liver failure, digestive malabsorption disease, being participating in an another clinical trial within the past 4 weeks, females that are pregnant or breastfeeding, or patients being judged to be unsuitable to be enrolled by the attending physician.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
(25(OH)D) | 3 months
  Change in serum 25-hydroxy vitamin D (25(OH)D) level

SECONDARY OUTCOMES:
serum sodium dismutase (SOD) | 3 months
  Change in serum sodium dismutase (SOD) levels
intact parathyroid hormone (iPTH) | 3 months
  Change in intact parathyroid hormone (iPTH) level
serum Malondialdehyde (MDA) | 3 months
  Change in serum Malondialdehyde (MDA) level
serum high sensitive C-reactive Protein (HsCRP) | 3 months
  Change in serum high sensitive C-reactive Protein (HsCRP) level
serum calcium level (Ca) | 3 months
  Change of serum calcium level (Ca),
serum phosphate level (PO4) | 3 months
  Change of serum phosphate level (PO4).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt